CLINICAL TRIAL: NCT03651258
Title: Facilitate the Transition From Passive Feeding to Active Feeding in Preterm Infants Through Early Play
Acronym: ALIJEU
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: ALIJEU
Record Dates: First submitted 2018-04-04; First posted 2018-08-29 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Immature Newborn; Feeding Behavior
Keywords: Feeding Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: patient who can benefit from the ALIJEU for certain meals
  Interventions: Behavioral: Implementation of ALIJEU
- Group of witnesses: patient who did not benefit from the ALIJEU

INTERVENTIONS:
Behavioral: Implementation of ALIJEU — The intervention concerns the passage from the passive feed (gastric tube) to the active feed (breast, feeding bottle).
  We propose to set up a pleasant moment just before his meal. This is a practical exercise of a few minutes.
  The aim of this special moment is to facilitate child-adult exchanges, improve active food intake and reduce the length of hospital stay.
  Groups: Experimental group

SUMMARY:
The approach described here is based both on theoretical concepts and on the work of several teams of researchers. By positioning the baby and the appropriate adult, a speech bath, a sustained look and an expressive face, it is hypothesized that this early communication exercise will significantly improve the transition from passive feeding, active feeding of the premature child, from a qualitative and quantitative point of view.

ELIGIBILITY:
Inclusion Criteria:

* Age of child at birth: <32 WA justified by the greater prevalence of oral disorders in these children.
* Age of the child at the start of the study: 35 WA, ie at the beginning of the establishment of active feeding within the unit.

Exclusion Criteria:

* Children with oral malformations
* Contra-indication to the realization to the ALIJEU (infection in progress, hemodynamic instability, etc.)
* Medical contraindications to oral diet

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Premate newborn with an age inferior to 32 weeks of amenorrhea at birth
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
age at the stoppage of enteral nutrition | 37 weeks of gestation

SECONDARY OUTCOMES:
Duration of feeding | 37 weeks of gestation
  Duration of the feeding in case of early game play
Quantities drunk | 37 weeks of gestation
  Evaluate the quantities drunk in case of early game play
Awakening | 37 weeks of gestation
  Duration of the the newborn's waking state at the time of suckling
Visual analogic scale for Satisfaction from 0 to 10 | 37 weeks of gestation
  Assessing the satisfaction of the ALIJEU practice for the mother and the care team

CONTACTS AND LOCATIONS:
Locations (1):
- CHI Créteil, Créteil, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No